IONA Consent form V4.0 12.04.2023 IRAS ID: 320784 Queen Mary Ethics of Research Committee Ref: QMERC22.170



## (IONA) Assessing the impact of non-tailpipe emissions from traffic on the asthmatic airway: Consent Form

Should you wish to participate in the study, please consider the following statements. Before signing the consent form, you should initial all or any of the statements that you agree with. Your signature confirms that you are willing to participate in this research, however you are reminded that you are free to withdraw your participation at any time.

| Statement | | initial box |
|---|---|---|
| 1. I confirm that I have read the Participant Information Sheet dated version for the above study; or it has been read to me. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | |
| 2. I understand that my participation is voluntary and that I am free to stop taking part in the study at any time without giving any reason and without my rights being affected. | | |
| 3. I understand that my data will be accessed by the research team. | | |
| 4. I understand that my data will be securely stored in Yvonne Carter Building, 58 Turner St,E1 2AB and in accordance with the data protection guidelines of the Queen Mary University of London for 25 years in pseudonymised form. | | |
| 5. I understand that I can access the information I have provided and request destruction of that information at any time prior open source publication. I understand that following open source publication. I will not be able to request withdrawal of the information I have provided. | | |
| 6. I understand that the researchers will not identify me in any publications and other study outputs using personal information obtained from this study. | | |
| 7. I confirm that samples and data collected can be used in the present study | | |
| 8. I confirm that samples can be used for DNA analysis. | | |
| 9. I confirm that samples collected can be stored in pseudonymised form in Sir Michael Uren Hub, Imperial College for future air pollution related research, subject to university research ethical approval. (Optional) | | |
| 10. I confirm that data collected can be stored in pseudonymised form in Yvonne Carter building, Queen Mary University London for future air pollution related research, subject to university research ethical approval. (Optional) | | |
| 11. I agree to take part in the above study. | | |
| Once completed, please return this signed forr records and a copy will be stored in our study i | m to Dr James Scales. A signed copy will be provided to y records. | ou for your |
| Participant name Date | Signature | |
| Name of researcher Date taking consent | Signature | e (whore |

I Dr James Scales confirm that I have carefully explained the nature, demands and any foreseeable risks (where applicable) of the proposed research to the participant and provided a copy of this form.

IONA Consent form: V4.0 12.04.2023





